CLINICAL TRIAL: NCT05542641
Title: T-mult: Exploring the Impact of TMS Induced Virtual Lesions on the Multimodal Brain Network and Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Linda Douw, Associate Professor, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NL82268.029.22
Record Dates: First submitted 2022-09-07; First posted 2022-09-15 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Healthy Cognition
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- real rTMS (Experimental): verum rTMS to the DLPFC, 1500 1Hz pulses at 120% RMT, 25 minutes total
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)
- sham rTMS (Sham Comparator): sham rTMS to the DLPFC, 1500 1Hz pulses at 120% RMT, 25 minutes total
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (rTMS) — real versus sham rTMS

SUMMARY:
T-mult is an experimental study using low-frequency (1Hz) single-sesson rTMS to the DLPFC (versus sham rTMS) to explore the effect of virtual lesions on the brain network and cognition in 100 healthy adults (20-65 years old).

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 65 years old
* Native Dutch speaker
* Able to provide written informed consent

Exclusion Criteria:

* History of diagnosed neurological or psychiatric disease (including traumatic head injury)
* Current and regular use of centrally acting drugs (recreational or prescribed, including analgesics), including the use of alcohol ~8 hours prior to an appointment
* Presence of any contraindications for MRI, MEG, or TMS (including resting motor threshold >75% of maximum stimulator output or no useful motor-evoked potential elicitable)
* Previous rTMS treatment

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
Cognitive change | baseline versus directly post-intervention (max. 8 weeks after baseline)
  Change in performance on a neuropsychological test measuring cognitive functioning in the domain of executive functioning

SECONDARY OUTCOMES:
Brain network change | baseline versus directly post-intervention (max. 8 weeks after baseline)
  Change in brain network organization as characterised by multimodal neuroimaging

CONTACTS AND LOCATIONS:
Overall Officials: Linda Douw, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Centers, location VUmc, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
In the pursuit of open science, we intend to make this dataset available to a larger part of the scientific community. Participants will be asked for their permission to do so in the Informed Consent form; if permission is given we will, upon completion of the study, upload coded data that has been scrubbed of all PHI (i.e. clear all PHI in the header information, deface MR images) to DANS (Data Archiving and Networked Services, www.dans.knaw.nl), a Dutch repository for research data. DANS allows for the use of a "restricted access" license for the reuse of data that ensures anyone who wishes to use the data acts in accordance with applicable local laws and regulations (e.g. AVG).
  Note that participants who are unwilling to provide permission to share their data will still be included in this study (their data will then not be uploaded to DANS).
Time Frame: Upon completion of the study
Access Criteria: See plan description